CLINICAL TRIAL: NCT01222364
Title: Delayed Cord Clamping in VLBW Infants Pilot Study
Brief Title: Delayed Cord Clamping in VLBW Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: William Oh, Lead Principal Investigator, Brown University, Women & Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0023; U10HD021364 (NIH); U01HD021438 (NIH); U10HD027853 (NIH); U10HD027904 (NIH); M01RR000080 (NIH); M01RR008084 (NIH)
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Cord Clamping (Active Comparator)
  Interventions: Procedure: Standard Cord Clamping
- Delayed Cord Clamping (Experimental)
  Interventions: Procedure: Delayed Cord Clamping

INTERVENTIONS:
Procedure: Standard Cord Clamping — Immediate clamping (<5 seconds) of the umbilical cord after delivery.
  Arms: Standard Cord Clamping
Procedure: Delayed Cord Clamping — Clamping of the umbilical cord at 30-45 seconds after birth.
  Arms: Delayed Cord Clamping

SUMMARY:
This study tested the feasibility of conducting a randomized controlled trial to vary the timing that doctors clamp the umbilical cord after birth in extremely low birthweight infants. The study also tested whether delaying cord clamping by 30-35 seconds and holding the newborn approximately 10 inches below the birth canal would result in increased hematocrit at 4 hours of age.

DETAILED DESCRIPTION:
This study tested the hypothesis that delaying clamping of the umbilical cord in extremely low birthweight (ELBW) infants would result in additional blood transfusion from the placenta to the baby, increasing the infant's blood volume and blood pressure. Higher blood pressure may improve blood flow to the brain that may reduce potential the risk of hypoxic ischemic encephalopathy (HIE) and/or intraventricular hemorrhage (IVH). The additional placental flow may also increase the amount of stem cells and cytokines flowing to the baby, improving immune status and reducing the risk of infection, while at the same time reducing the need for blood transfusions in the neonatal period.

This was a pilot study to test the feasibility of having obstetricians delay cord clamping for 30-45 seconds, and to confirm whether the procedure significantly increases the baby's hematocrit during the first 4 hours of life.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at participating centers at 24-27 weeks gestation
* Singletons
* Obstetrician approval for enrollment
* Parental consent

Exclusion Criteria:

* Prenatally diagnosed major congenital anomalies
* Intent to withhold or withdraw care
* Significant bleeding due to placenta previa or abruption

Max Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2000-06; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Infants enrolled | 6 months
  Number of infants enrolled in the pilot within 6 months.

SECONDARY OUTCOMES:
Intention to treat | 6 months
  Identify obstetricians willing to participate in randomizing subjects.
Hematocrit level | 4 hours of age
Arterial blood pressure | 12 hours of age
Use of volume expansion or pressor therapy | 24 hours of age
Blood transfusions | Until hospital discharge or 120 days of life

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island

REFERENCES:
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/